CLINICAL TRIAL: NCT06765772
Title: Combined Ultrasound Guided Bilateral Rectus Sheath and Erector Spinae Plain Blocks Versus Erector Spinae Plain Block for Intra and Postoperative Analgesia in Elective Abdominoplastic Surgeries. a Randomized Controlled Double Blinded Trial.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hassan Mohamed Ali, Professor of Anesthesia, Cairo University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: MS-370-2024
Record Dates: First submitted 2024-12-28; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-12

CONDITIONS: Abdominoplasty; Perioperative Analgesia
Keywords: Rectus sheath block; Erector spinae plane block

STUDY DESIGN:
Intervention Model Description: 2 groups A&B In Group A: GA along with combined Rectus sheath and Erector spinae plane blocks. In Group B: General anesthesia along with Erector spinae plane block alone.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Active Comparator): 20 Adult patients scheduled for elective abdominoplastic surgeries under general anethesia
  Interventions: Procedure: Erector spinae plane block; Procedure: Rectus sheath block
- Group B (Active Comparator): 20 Adult patients scheduled for elective abdominoplastic surgeries under general anethesia
  Interventions: Procedure: Erector spinae plane block

INTERVENTIONS:
Procedure: Erector spinae plane block — the patient will recieve ultrasound guided erector spinae plane blockbe. A 20-gauge needle will be placed between the erector spinae muscle and the thoracic transverse processes at the level of T10 using an 'in plane' technique, 20 ml of (0.25% bupivacaine and 1% xylocaine) will be injected on each side.
Procedure: Rectus sheath block — the patient will recieve ultrasound guided rectus sheath block. An 18-gauge needle will be introduced- in plane- just below the costal margin at an angle of approximately 45 degrees to the skin between the rectus abdominis muscle and posterior rectus sheath. 10 ml of (0.25% bupivacaine and 1% xylocaine) will be injected on each side.
  Arms: Group A

SUMMARY:
The goal of this clinical trail is to determine if bilateral erector spinae plane block alone can provide good perioperative analgesia for abdominoplastic surgery patients or it is better to give combined bilateral rectus sheath and erector spinae plane blocks to achieve effective intraoperative and postoperative analgesia with minimal morphine consumption in such operations in which there is an extensive surgical dissection and a high risk of respiratory problems.

DETAILED DESCRIPTION:
This study is randomized controlled trail in which 40 adult patients (male or female) scheduled for elective abdominoplastic surgeries during the study duration will be randomized into to equal groups to investigate the efficacy of erector spinae plane block alone versus the efficacy of combine use of erector spinae and rectus sheath plane block for intra and postoperative analgesia in abdominoplastic surgery patients.

ELIGIBILITY:
Inclusion Criteria:

* patients Age from 21 to 60 years ,Male and female patients ,ASA I, II patients scheduled for elective abdominoplastic surgeries during the study duration.

Exclusion Criteria:

* Patient refusal, Age less than 21 and above 60 years old, ASA III, IV patients., Infection at the site of injection, Opioid addiction, Allergy to any used substances (lidocaine, bupivacaine)., Preexisting severe or uncontrolled respiratory, renal or cardiac disease. , INR more than 1.5 and platelets less than 100000.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Primary outcome | one hour
  Visual Analogue Scale (VAS) measures pain intenesity one hour after extubation

SECONDARY OUTCOMES:
Secondary Outcome | first 24 hours postoperative
  Total morphine consumption during 1st 24 hours postoperatively
Secondary Outcome | During opration
  Total intraoperative fentanyl consumption.

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Mohamed Ali, Phd, Study Director — Professor of anesthesia Cairo university faculty of medicine
Locations (1):
- Cairo university hospital, Cairo, Cairo Governorate, Egypt